CLINICAL TRIAL: NCT03562988
Title: A Randomized, Examiner-blind, Comparator-controlled, Cross-over Bioequivalence Study on Vitamin C in Healthy Adults
Brief Title: Bioequivalence Study on Vitamin C in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ST-7666
Record Dates: First submitted 2018-05-02; First posted 2018-06-20 (Actual); Results first posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-04

CONDITIONS: Dietary Exposure
Keywords: Measure Absorption of Vitamin C in Blood
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C gummy, Then Vitamin C Caplet (Other): The study consisted of two single-day study periods separated by a 7-day washout. At the first study day, a single oral dose of vitamin C gummy (1007.2mg) was orally administered following a 12 hour fasting period. After a 7 day washout period, a single oral dose of vitamin C caplet (1027.9mg) was orally administered following a 12 hour fasting period.
  Interventions: Dietary Supplement: Vitamin C gummy; Dietary Supplement: Vitamin C tablet
- Vitamin C tablet, Then Vitamin C gummy (Other): The study consisted of two single-day study periods separated by a 7-day washout. At the first study day, a single oral dose of vitamin C caplet (1027.9mg) was orally administered following a 12 hour fasting period. After a 7 day washout period, a single oral dose of vitamin C gummy (1007.2mg) was orally administered following a 12 hour fasting period.
  Interventions: Dietary Supplement: Vitamin C gummy; Dietary Supplement: Vitamin C tablet

INTERVENTIONS:
Dietary Supplement: Vitamin C gummy — vitamin C
Dietary Supplement: Vitamin C tablet — vitamin C

SUMMARY:
The objective of this exploratory pharmacokinetic research study is to demonstrate that both caplets and gummies provide an effective dose of ascorbic acid in healthy adults.

DETAILED DESCRIPTION:
This randomized, examiner-blind, cross-over study evaluates the bioequivalence of a gummy containing vitamin C relative to a caplet comparator product in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 to 29.9 kg/m2 (+/- 1 kg/m2)
* Healthy as determined by laboratory results and medical history
* Maintains current level of physical activity throughout duration of study
* Does not donate blood for the next 3 months after completing study
* Avoidance of foods and beverages fortified with vitamin C for at least 7 days prior to enrollment and duration of study
* Avoidance of citrus foods, citrus juices, and tomato juice for at least 7 days prior to enrollment and duration of study
* Non smoker or ex-smoker > 1 year
* Has given voluntary, written informed consent to participate in study
* Agrees to avoid high caffeine and alcohol intake 72 hours prior to in-clinic test days and during the 24-hour in-clinic test days
* Females not of child bearing potential, defined as having had a hysterectomy, oophorectomy, bilateral tubal ligation or are post-menopausal
* Females of child bearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods include hormonal contraceptives, double-barrier method, intrauterine devices, non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s) and/or vasectomy of partner

Exclusion Criteria:

* Women who are pregnant, breast feeding, or planning to become pregnant during the trial
* Duodenal or gastric ulcer, gastritis, hiatus hernia, or GERD within past 3 months
* History of irritable bowel syndrome and related disorders
* Significant gastrointestinal disease (includes but not limited to Celiac disease)
* History of malabsorption
* Unstable medical conditions as determined by the Qualified Investigator
* Blood pressure greater than 150/90 mmHg
* Cancer except skin cancers completely excised with no chemotherapy or radiation following and with a negative follow up. (Volunteers with cancer in full remission for more than 4 years after diagnosis are acceptable)
* Clinically significant abnormal laboratory results at screening
* Metabolic disease or chronic diseases (ex/ hyperlipidemia, hypertension, hypercholesterolemia)
* Type I or Type II diabetes
* History of kidney stones
* Use of prescription or over the counter products known to interact with vitamin C within 72 hours of enrollment and duration of trial such as aspirin and NSAIDs, aluminum, iron, and proton pump inhibitors
* Use of acute over the counter medication within 72 hours of test product dosing
* Use of tobacco products within the last year
* More than 2 alcoholic drinks per day
* Drug abuse within 1 year of enrollment
* Use of medicinal marijuana
* Immunocompromised individuals such as individuals that have undergone organ transplantation or individuals diagnosed with HIV
* Individuals who have planned surgery during the course of the trial
* St. John's wort in the last 30 days prior to enrollment and duration of study
* Use of vitamin C, multivitamins containing vitamin C, or foods or beverages fortified with vitamin C and other natural healthy products containing vitamin C within 7 days of enrollment and duration of study
* Consumption of citrus foods, citrus juices, and tomato juice with 7 days of enrollment and duration of study
* Use of anticoagulants, barbiturates, tetracycline antibiotics, beta-blockers, cyclosporine, prednisone, tricyclic antidepressants, diuretics and nitrate medications
* Use of natural health products/dietary supplements with 7 days of enrollment or duration of study
* Current diagnosis and history of blood/bleeding disorders
* Current diagnosis and history of anemia of any etiology defined as hemoglobin < 145 g/L for males and < 123 g/L for females
* History of hemoglobinopathies such as sickle cell anemia or thalassemia, sideroblastic anemia
* History of hemochromatosis
* Blood donation in the past 3 months
* Individuals who plan to donate blood during the study or within 30 days of completing the study
* Participation in a clinical research trial within 30 days prior to enrollment
* Allergy or sensitivity to supplement ingredients or to any food or beverage provided during the study
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Qualified Investigator's opinion nay adversely affect an individual's ability to complete the study or its measures or which may pose significant risk to the individual

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annahita Ghassemi, Study Director — Church & Dwight Company, Inc.
Locations (1):
- Church & Dwight Co., Inc., Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evans M, Guthrie N, Zhang HK, Hooper W, Wong A, Ghassemi A. Vitamin C Bioequivalence from Gummy and Caplet Sources in Healthy Adults: A Randomized-Controlled Trial. J Am Coll Nutr. 2020 Jul;39(5):422-431. doi: 10.1080/07315724.2019.1684398. Epub 2019 Nov 20. PMID 31747355

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cross over study. Participants received each treatment at one of the two treatment visits.
Period: Overall Study
Arm/Group | Vitamin C Gummy, Then Vitamin C Caplet | Vitamin C Tablet, Then Vitamin C Gummy
Started | 17 | 18
Completed | 15 | 15
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Population: Cross over study. Participants randomly received one treatment at one of the two dosing days and the other treatment at the second dosing day.
Groups:
- All Study Participants: All Study Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Plasma L-ascorbic Acid as Total Area Under the Curve [AUC(0-24 Hours)]
Description: Mean Plasma L-ascorbic Acid as Total Area Under the Curve [AUC(0-24 hours)]
Time Frame: baseline, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours
Population: Includes all Participants from treatment day 1, including those did not participate in treatment day 2.
Measure: Mean (Standard Deviation); unit: μmol*min/L
Groups:
- Vitamin C Gummy: A single oral dose of vitamin C gummy
- Vitamin C Caplet: A single oral dose of vitamin C caplet
Arm/Group | Vitamin C Gummy | Vitamin C Caplet
Number analyzed (Participants) | 32 | 33
μmol*min/L | 1114.66 (236.81) | 1149.09 (237.89)

2. Primary Outcome: Mean Leukocyte L-ascorbic Acid as Total Area Under the Curve [AUC(0-24 Hours)]
Description: Mean Leukocyte L-ascorbic Acid as Total Area Under the Curve [AUC(0-24 hours)] for All Study Participants
Time Frame: baseline, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours
Population: Includes all Participants from treatment day 1, including those did not participate in treatment day 2.
Measure: Mean (Standard Deviation); unit: nmol*min/10^8 leukocytes
Groups:
- Vitamin C Gummy: A single oral dose of vitamin C gummy to monitor vitamin C blood levels
  Vitamin C gummy: vitamin C
- Vitamin C Tablet: A single oral dose of vitamin C tablet to monitor vitamin C blood levels
  vitamin C tablet: vitamin C
Arm/Group | Vitamin C Gummy | Vitamin C Tablet
Number analyzed (Participants) | 32 | 33
nmol*min/10^8 leukocytes | 273.20 (115.70) | 297.20 (105.86)

3. Primary Outcome: Mean Plasma L-ascorbic Acid as Cmax
Description: Mean Plasma L-ascorbic Acid as Cmax
Time Frame: baseline, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours
Population: Includes all Participants from treatment day 1, including that those did not participate in treatment day 2.
Measure: Mean (Standard Deviation); unit: μmol/L
Groups:
- Vitamin C Gummy: A single oral dose of gummy vitamin C to monitor vitamin C blood levels
  Vitamin C gummy: vitamin C
- Vitamin C Tablet: A single oral dose of tablet vitamin C to monitor vitamin C blood levels
  Vitamin C tablet: vitamin C
Arm/Group | Vitamin C Gummy | Vitamin C Tablet
Number analyzed (Participants) | 32 | 33
μmol/L | 72.75 (15.74) | 78.97 (20.51)

4. Primary Outcome: Mean Leukocyte L-ascorbic Acid as Cmax
Description: Mean Leukocyte L-ascorbic Acid as Cmax
Time Frame: baseline, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours
Population: Includes all Participants from treatment day 1, including those did not participate in treatment day 2.
Measure: Mean (Standard Deviation); unit: nmol/10^8 leukocytes
Arm/Group | Vitamin C Gummy | Vitamin C Tablet
Number analyzed (Participants) | 32 | 33
nmol/10^8 leukocytes | 22.96 (18.91) | 22.74 (13.98)

5. Secondary Outcome: Mean Plasma Vitamin C Absorption Rate as Tmax
Description: Mean Time of maximum Vitamin C concentration
Time Frame: baseline, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours
Population: Includes all Participants from treatment day 1, including those did not participate in treatment day 2.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vitamin C Gummy | Vitamin C Tablet
Number analyzed (Participants) | 32 | 33
hours | 2.59 (0.71) | 2.88 (1.11)

6. Secondary Outcome: Mean Leucocyte Vitamin C Absorption Rate as Tmax
Description: Mean Time of maximum Vitamin C concentration
Time Frame: baseline, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours
Population: Includes all Participants from treatment day 1, including those did not participate in treatment day 2.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vitamin C Gummy | Vitamin C Tablet
Number analyzed (Participants) | 32 | 33
hours | 6.73 (3.61) | 4.58 (3.84)

ADVERSE EVENTS:
Time Frame: Participants entered any AE's in a daily diary from the initiation of the study until 24 hours after the last oral dosing. Additionally, participants were asked about AE's at each visit.
Arm/Group | Vitamin C Gummy | Vitamin C Tablet
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 2/32 | 1/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin C Gummy (N=32) | Vitamin C Tablet (N=33)
Abnormal Neutrophil Count (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Mild Somnolence (General disorders) | 1 (1) | 0 (0)
Mild Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality and Master Service Agreement

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03562988/Prot_SAP_000.pdf